Study Identifiers: DI SLE. Auto 2003; NCT 00278538

<u>Study Title</u>: Cyclophosphamide and Rabbit Antithymocyte Globulin (rATG)/Rituximab in Patients with Systemic Lupus Erythematosus

# Cyclophosphamide and rATG/rituximab in Patients with Systemic Lupus Erythematosus: Phase II Trial

# FDA sponsor and Principal Investigator:

Richard Burt, MD
Division of Immunotherapy
Northwestern University Medical Center
E-mail: rburt@northwestern.edu

# Co-Investigators:

Eric Ruderman, M.D.
Division of Rheumatology
Northwestern University and Northwestern Memorial Hospital

Kathleen Quigley, R.N., M.B.A. Northwestern University

Kimberly Yaung, RN Northwestern Medical Faculty Foundation

#### Statistician:

Borko Jovanovic, M.S., Ph.D. Northwestern University

# Cyclophosphamide and rATG/rituximab in Patients with Systemic Lupus Erythematosus: Phase I Trial

#### STUDY SYNOPSIS

**Participating Sites:** 

Northwestern Memorial Hospital

Accrual Objective:

40 participants

Primary Study Objective:

The primary efficacy outcome is overall survival and the proportion of participants who achieve and maintain remission after transplant. Remission is defined according to the RIFLE as duration on no immune suppressive medications except

physiologic doses of prednisone (<10 mg/day) or corticosteroid equivalent and or hydroxychloroquine.

**Trial Treatment:** 

Participants will receive high dose cyclophosphamide (200 mg/kg), rATG (6mg/kg) and rituximab 200mg, followed by

rescue with peripheral stem cells.

**Study Duration:** 

The trial duration will be 5 years.

**Study Population:** 

Participants with systemic lupus erythematosus (SLE) will be enrolled in the study. Participants must be 16 to 60 years of age and must meet at least 4 of 11 American College of Rheumatology (ACR) classification criteria for SLE.

# 1. Background Information and Scientific Rationale

#### 1.1. Background Information on Systemic Lupus Erythematosus

Systemic lupus erythematosus (SLE) is a multi-system, inflammatory disorder characterized by the production of antibodies that react with many different self-antigens. Despite differences in presentation, manifestations, and clinical course, the common factor for patients with systemic lupus erythematosus (SLE) is hyper-reactivity of T and B cells to endogenous stimuli.

Currently, in developed countries, mortality from SLE is estimated at 3 per million person-years. A number of factors are associated with poor prognosis; these include the presence of renal disease causing an elevation in serum creatinine or urine protein excretion above normal, hypertension, diffuse proliferative glomerulonephritis on renal biopsy, chronic changes on biopsy, lung involvement, a high Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score at the time of first lupus clinic visit, anemia, thrombocytopenia, and antibodies to phospholipids. 1

Rose's criteria for proof that a disease is autoimmune requires transfer of disease to a person by transfer of antibodies or immune cells from an afflicted individual.3 Evidence of a suspected autoimmune etiology for most diseases is indirect and based on laboratory evidence of immune responses to self that are quantitatively and/or qualitatively different from a healthy population, and response to anti-inflammatory and/or immunosuppressive therapies. The autoimmune nature of SLE is supported by several observations. First, nephritis may be induced in asymptomatic mice by injection of anti-DNA antibody from mice afflicted by a lupus-like nephritis4 and occurs in normal mice made transgenic for the heavy and light chains of an IgG antibody to double-stranded DNA.5 Second, in SCID mice that cannot reject xenogeneic proteins, injection of anti-DNA antibody from patients with SLE induces proteinuria.<sup>6</sup> Third, in 1959. healthy individuals were transfused with 300 mls of plasma from LE positive patients with SLE.7 There was no observable clinical effect, but the patients developed transient LE cells, which result from phagocytosis of antibody coated nuclei. It is unknown if continued transfusions of SLE plasma could have precipitated clinical disease. Fourth, disease activity for most patients with SLE correlates with serum levels of anti-double stranded DNA (anti-ds DNA) antibody titer.<sup>8</sup> In general, SLE is responsive to immune suppression, indirectly supporting an autoimmune pathogenesis.

#### 1.2. Clinical Classification of Disease Staging

Multiple indices exist to measure or characterize disease activity. Activity instruments include the British Isles Lupus Assessment Group scale (BILAG),<sup>9</sup> Systemic Lupus Erythematosus Disease Activity Index (SLEDAI),<sup>10</sup> Systemic Lupus Activity Measure (SLAM),<sup>11</sup> and the Lupus Activity Index (LAI).<sup>12</sup> The instrument employed depends on institutional and investigator familiarity.

# 1.3. Underlying Immunologic Mechanisms

SLE is probably a genetically heterogeneous disease influenced by multiple loci. In New Zealand Black / New Zealand White F1 hybrids (NZB/NZW) mice, various mating crosses of lupus prone mice, as well as backcrosses to normal mice have linked murine lupus to 38 different genomic loci. Depending upon the crossmating strains, different loci with different nomenclature have been identified. Examples of nomenclature for loci associated with SLE are: Lrdm (lpr renal disease modifier), nba (New Zealand Black autoimmunity), Lbw (lupus NZB x NZW), and Sle (systemic lupus erythematosus). Murine lupus-like disease is polygeneic with multiple genes (including Sle1, Sle3, Ldrm1, Ldrm2, nba1, nba2, Lbw3) contributing. Some loci are associated with one or more of the following: glomerulonephritis, vasculitis, anti-ds DNA, anti-chromatin antibody, lymphoproliferation, or splenomegaly.

No single gene is sufficient to cause disease in animal studies. This suggests that human SLE is also polygeneic with multiple potential combinations predisposing to SLE. Genetic analysis predicts that many genes are involved in the expression of lupus in humans.<sup>23</sup> Class II molecules, DR2 and DR3, have been associated with lupus in North American whites. Various combinations of SLE-prone genes among different patients may explain why patients with SLE can have highly variable organ involvement and clinical symptoms.

Additionally, it is believed that genetic disposition alone is not sufficient to induce lupus in humans. In monozygotic twins, 30-50% are concordant for disease.<sup>24</sup> The disease is much more common in females than males, with approximately 7:1 ratio of women to men in child-bearing years.<sup>25</sup> A multi-factorial etiology including genetic predisposition, permissive sex hormone status, and environmental interaction are probably necessary for development of clinical disease.

The common thread in disease pathogenesis in humans is T and B cell hyperreactivity. T cells from patients with SLE provide help to B cells to produce autoantibodies.<sup>26</sup> An unaffected person's peripheral T cells are less than 1% positive for CD69 (a marker of activation), and upon ex vivo exposure to a mitogen such as PMA (4Bal Phorbol 12 Myristrate 13 Acetate) more than 80% of the T cells will present CD69 within 4-6 hours. Pretransplant T cells from patients with lupus display the activation marker CD69 in 10-54% of the unstimulated cells and fail to appropriately further upregulate CD69 expression in response to PMA.27 Fresh T cells and T cell lines from patients with lupus display enhanced TCR-mediated protein tyrosine phosphorylation and intracellular free calcium concentrations. 28,29 Therefore, T cells from patients with lupus may "overshoot" surface mediated signaling events. This is further supported by the observation that expression of second signal molecules such as CD40 ligand are increased on the T cells and B cells of patients with SLE 30 and levels of soluble CD40L are increased in sera.31 Lymphocytes from some patients with active lupus also display a Th2 cytokine skewing.32 In general, Th2

cytokines promote B cell antibody production. The pattern of cytokine expression in SLE cells and patient sera is complex and multiple studies have yielded different results, depending on methods used and characteristics of patients studied.<sup>33</sup> There is general agreement that levels of IL-10 are increased in sera of many patients, and generation of TGF-beta by PBL is significantly lower compared to normal individuals.<sup>34</sup>

The pretransplant T cell receptor CDR3 repertoires are also skewed indicating expansion of reactive T cells.<sup>35</sup> After transplant, these pretransplant T cell hyperactivation abnormalities normalize.<sup>27</sup> Although encouraging, the post-transplant duration of a normalized T cell phenotype is unknown. Analysis of B cell activation, signal transduction and immunoglobulin receptor skewing is yet to be performed on the pre and post-transplant samples.

It appears that T cell stimulation of B cells occurs in the pathogenesis of lupus patients. Once stimulation of B-cells has taken place and anti-self immunity has been stimulated, the memory for anti-self immune responses is retained and reactivation of pathogenic antibodies occurs with greater ease in subsequent relapses.

### 1.4. Current Therapy

Mortality from SLE has markedly improved due to more aggressive antiinflammatory and immunosuppressive treatments as well as improved supportive care from dialysis, apheresis, and newer anti-hypertensive and antibiotic medications. For patients with diffuse proliferative glomerulonephritis, 5-year survival in the 1950's was almost zero percent. 28 With introduction of high-dose corticosteroids in the 1960's, the 5-year survival for this subset improved to 25%.38 Following addition of oral cyclophosphamide and azathioprine, 5-year survival in severe lupus nephritis improved to 40-70%. In the 1980's, introduction of intravenous pulse cyclophosphamide (500-1000 mg/m² monthly for six months and then every three months for six months) improved 5-year survival to 80%.29 More recent therapies for SLE include cyclosporine and mycophenolate mofetil.40 Twelve-month survival rates and response rates were similar in patients with lupus nephritis (approximately 80%) treated with either daily oral cyclophosphamide for 6 months (followed by daily oral azathioprine for 6 months) compared to mycophenolate mofetil daily for 12 months. The current standard of care in the USA for patients with SLE nephritis that is life-threatening is intravenous pulse cyclophosphamide (500-1000 mg/m²) per month for six months and then every three months for six months. Despite these advances for high risk SLE, mortality is 20% at 2 years and 35% at 5 years which is an unacceptably high mortality for predominately young women between ages 20 to 30.



# 1.5. A Summary of Preclinical and Clinical Experience

# 1.5.1. Preclinical experience with hematopoietic stem cell transplantation

Animal autoimmune diseases that are induced by immunization with adjuvant or self-peptide and adjuvant may be ameliorated by syngeneic or pseudoautologous hematopoietic stem cell transplantation (HSCT).41-52 Immunization with adjuvant and either myelin basic protein (MBP) or proteolipid protein (PLP) peptides induces a T cell mediated demyelinating disease, Experimental Autoimmune Encephalitis (EAE). Depending upon the animal model. EAE may be similar to multiple sclerosis (MS) -- monophasic, relapsing-remitting with secondary progression or progressive from onset. In particular, EAE in Swiss Jackson Laboratory/Jackson (SJL/J) mice is a relapsing remitting and secondarily progressive disease. Several investigators have demonstrated a cure, decreased relapse rates, or decreased disease severity in SJL/J mice undergoing syngeneic HSCT. 43,45,49,50 Some investigators have reported post transplant antigen specific tolerance suggesting that the HSCT induced tolerance through clonal deletion or anergy of myelin reactive cells.<sup>43</sup> Other laboratories have reported clinical and histologic remission after syngeneic HSCT but persistence of myelin reactive T cells post transplant.<sup>45</sup> This would suggest that the mechanism of clinical tolerance might be through a cytokine shift, enhancement of regulatory cells, or inability of T cells to home to the central nervous system (CNS).

Due to the expense of long term animal housing, most EAE experiments are performed prior to disease onset in order to abort disease initiation or shortly after disease onset in order to ameliorate its course. It is unlikely that such experiments are applicable to patients with a long duration of MS with

accumulated disease burden and tissue damage. Syngeneic HSCT performed in mice with chronic EAE, unlike the results in acute EAE, failed to demonstrate neurologic improvement.<sup>45</sup> Histologic analysis revealed chronic scarring with glial proliferation that is unaffected by HSCT.<sup>45</sup> To be effective as therapy for EAE, it is hypothesized that HSCT needs to be performed early in disease course during its inflammatory stage and before accumulation of disease burden.

Murine bone marrow transplants are performed by euthanizing and removing the femur from the donor and using a syringe to flush out the marrow cells. It is technically difficult and inhumane to perform a murine autologous transplant since the surviving recipient's legs would have to be amoutated. However, marrow could be harvested from a syngeneic donor in the same active stage of EAE as the recipient; this is referred to as a pseudo autologous transplant. HSCT of EAE using pseudo autologous donors suggests that infused lymphocytes contaminating the graft may contribute to relapse. 46 This indicates that lymphocyte depletion of grafts may be important in decreasing post transplant relapse following autologous HSCT. Several other environmentally induced animal autoimmune diseases are improved or cured by syngeneic or autologous HSCT. These include experimental autoimmune myasthenia gravis<sup>52</sup> and adjuvant- and collageninduced arthritis. 42,44 In a mouse model of lupus-like autoimmunity accompanied by coronary artery disease (associated with antibodies to phospholipid), transplantation of syngeneic stem cells depleted of T cells prevents disease. 53 Nephritis can also be prevented in BXSB lupus mice with establishment of mixed chimerism using bone marrow cells.<sup>54</sup> However. murine models of lupus are stem cell defects that require an allogeneic transplant to be cured.

A spontaneous lupus-like illness occurs in many species including dogs, monkeys, and mice. Most studies have, for economical reasons, been confined to highly inbred murine strains.55 New Zealand Black (NZB) mice develop a spontaneous hemolytic anemia. When NZB mice are mated to normal New Zealand White (NZW) mice the F1 offspring (NZB x NZW) or B/W mice develop antinuclear antibodies (ANA), anti-ds DNA antibodies, and early death from glomerulonephritis.58 Disease occurs in both males and females but is more severe in females. The B/W lupus-like illness arises from polygenic loci contributed by both parents. At least 8 genes on multiple chromosomes are involved and may be inherited in a dominant or recessive manner.<sup>57</sup> Individual loci appear to be linked to different stages of disease (e.g. antibody formation, glomerulonephritis, or mortality). Mating NZB mice to another normal mouse strain (SWR) also results in offspring (SNF1) with a lupus-like illness. SNF1 mice have disease similar to B/W mice manifest by spontaneous onset autoantibodies, glomerulonephritis, female predominance. and linkage to polygenic loci.58

The Murthy Roth lab lymphoproliferative (MRL/lpr) mouse develops massive lymphadenopathy, glomerulonephritis, erosive arthritis, polyarteritis, hypocomplementemia, and a variety of autoantibodies including: ANA, anti-ds DNA, anti-Sm, rheumatoid factor, and anti-phospholipid antibodies.<sup>59</sup> The congenic MRL/+/+ mouse develops similar serologic abnormalities and glomerulonephritis but does not develop lymphoproliferation and disease is milder with a life span of up to 24 months. In contrast, MRL/lpr mice die within 3-6 months. As mentioned, MRL/lpr and MRL/+/+ mice are congenic which means that they have been bred for consecutive generations to differ in only one loci. This single loci difference, the lpr gene, encodes a defective Fas molecule.<sup>60</sup> Surface Fas expression, when engaged by the Fas ligand, induces apoptosis. Therefore, a single gene defect, Fas, results in an accelerated autoimmune phenotype in a genetically susceptible strain.

The BXSB strain of mice also develops a spontaneous lupus-like illness.<sup>61</sup> The disease is worse in males than females. Acceleration of disease phenotype in males is due to a Y chromosome gene termed Y chromosome autoimmune accelerator (*Yaa*).<sup>62</sup> The function of the *Yaa* gene is unknown but unless expressed in a susceptible strain is unable to cause disease. *Yaa* has been postulated to increase expression of adhesion molecules aiding T cell stimulation of B cells. Finally, male offspring of BXSB x NZW mice develop antibodies to DNA, platelets and phospholipids and die of accelerated coronary artery disease.<sup>63</sup> This is pertinent to lupus patients since some suffer from increased vascular events including coronary artery disease.

Immune cells arise from the hematopoietic compartment. Therefore, hematopoietic (i.e. bone marrow) transplantation from a non-disease susceptible donor has been attempted to treat animal autoimmune disease. Allogeneic bone marrow transplantation (i.e. immune ablation and infusion of hematopoietic stem cells from a normal strain) prevents and/or cures lupus-like disease in BXSB and B/W mice. While allogeneic HSCT can cure lupus-like disease, it is generally thought that autologous or syngeneic marrow transplantation would transplant disease prone cells and be ineffective. Although not curative, lymphocyte depleted syngeneic marrow transplantation induces life-prolonging remissions in MRL/Ipr mice.

Application of these murine lupus-like models to SLE must be done with caution since the mice originate from highly inbred strains. Murine models are important to identify genetic loci mediating autoimmune phenomena. However, in outbred human populations, environmental exposure and regulatory cells and other suppressor mechanisms may have significant roles in controlling disease-associated genes. In fact, unlike murine models of lupus, patients with SLE can enter spontaneous remissions off therapy. Therefore, the potential for autologous HSCT to cure SLE remains possible but uncertain.

# 1.5.2. Preliminary clinical experience with hematopoietic stem cell transplantation

Anecdotal case reports of patients with a coincidental autoimmune disease and a malignancy provide further support and rationale for trial design. Refractory autoimmune diseases enter remission sometimes for several years. In these anecdotal reports, the indication for transplant was a malignancy or aplastic anemia and the outcome reported retrospectively, and therefore in most cases a detailed pre transplant evaluation by a rheumatologist or neurologist is missing. The results in these cases are that the autografts were usually not purged of lymphocytes, and the transplants were not tailored as therapy for an autoimmune disease. Duration of response appeared shorter for rheumatoid arthritis compared to systemic lupus erythematosus. Too few patients have been reported for other autoimmune diseases and long-term results of response to treatment in those that relapse as well as duration of remission in those that had not relapsed remains unknown.

Autologous transplantation performed for malignant disease is associated with a prolonged, post transplant "immunosuppressive" phenotype, which has recently been reported by our group to exist after autologous transplantation of autoimmune diseases as well. This generalized "suppresser" phenotype is manifest by a low CD4 count, elevated CD8 percentage, an inverted CD4/CD8 ratio, and an early predominance of CD45RO memory cells followed after 3-6 months by recurrence of CD45RA naive cells. There is speculation that high dose immunosuppression, by inducing apoptosis of disease causing lymphocytes and imposing a post transplant suppresser phenotype, may be beneficial in inducing a sustained remission of lupus. We, therefore, chose the safer autologous stem cells over an allogeneic source of stem cells for the phase I study.

#### 1.5.3. Phase I study at Northwestern University

A phase I study to perform lymphocyte depleted autologous hematopoietic stem cell transplantation for patients with poor prognosis systemic lupus erythematosus was initiated in 1996 following U.S. FDA approval. Thirty-one patients have undergone transplant. We reported the first patient as a letter to the *New England Journal of Medicine*<sup>80</sup> and subsequently reported further results as articles in *The Lancel*<sup>35</sup> and *Arthritis and Rheumatism*<sup>36</sup>. The reasoning that went into the development of that protocol is recounted here as it is relevant to our current proposal. Cyclophosphamide was chosen as the immunosuppressive regimen because of its established effectiveness at conventional dosage in the treatment of lupus. All transplant candidates had to have failed monthly pulse cyclophosphamide at 500-1000 mg/m². We recognized that the dose limiting toxicity of cyclophosphamide, unlike most

alkylating agents, is not hematopoietic. Even without reinfusion of stem cells, cyclophosphamide-induced cytopenias will resolve. In recognition of this fact, some investigators have performed immunosuppressive trials in autoimmune diseases using high dose cyclophosphamide without stem cell reinfusion. We chose to reinfuse G-CSF mobilized hematopoietic stem cells in order to minimize the duration of cyclophosphamide induced neutropenia. We reasoned that the patients who met our eligibility criteria, having been heavily pretreated with immunosuppressive medications, would be at high risk of opportunistic infection. This proved true. Two patients who met our eligibility criteria could not be taken to transplant because of opportunistic infections (cytomegalovirus pneumonitis and mucormycosis). Both were diagnosed prior to transplantation and after a transient period of neutropenia (ANC < 500/ul for 2-3 days) associated with stem cell mobilization.

#### Methods

Method of Harvesting Stem Cells: Hematopoietic stem cells were mobilized with cyclophosphamide (2 g/m²) and G-CSF. Engraftment kinetics is faster with G-CSF mobilized peripheral blood stem cells compared to marrow. Due to the anticipated high risk of infection in patients with SLE, we felt that the rapid engraftment of peripheral blood stem cells would be superior to that of marrow. In fact, most autologous transplants for malignancies now use peripheral blood mobilized stem cells rather than marrow due to more rapid engraftment, less infections, and more rapid hospital discharge. We were concerned that attempts to mobilize peripheral blood stem cells with G-CSF (an inflammatory cytokine) would be dangerous for patients with active SLE. For this reason, cyclophosphamide (2.0 mg/m²) was given first with G-CSF started 4-5 days later. This dose of cyclophosphamide caused neutropenia of 1-3 days duration. Leukapheresis was initiated when the post nadir white blood cell count reached more than 1,000/ul (1.0 x 109/liter). Daily apheresis was continued until the number of harvested progenitor cells reached a minimum of 1.4 x 10<sup>8</sup> CD34<sup>+</sup> cells/kg body weight after selection. The mobilized peripheral blood stem cells were lymphocyte depleted via selection for CD34 positive cells using the CEPRATE SC Stem Cell Concentrator (CellPro, Bothell, Washington).

Patient selection: In order to select for patients at high risk for early mortality, we chose patients with active visceral disease despite the use of pulse cyclophosphamide and corticosteroids. Cyclophosphamide must have been given for at least 6 months for patients with nephritis (WHO class III or class IV glomerulonephritis). With other visceral organ involvement, failure to prevent life-threatening manifestations (e.g. cerebritis, transverse myelitis, pulmonary hemorrhage, restrictive lung disease or cardiac failure) between pulses of cyclophosphamide was also an indication.

Conditioning Regimen: On pre-transplantation days –5 to –2, patients were given daily intravenous doses of 50mg/kg cyclophosphamide. On pre-transplantation days –4 to –2, patients were given 250-1000 mg methylprednisolone intravenously, followed by 30 mg/kg antithymocyte globulin.

Upon admission to the HEPA-filtered hematology/oncology floor, patients started a low microbial diet which was discontinued when the absolute neutrophil count rebounded to  $0.5 \times 10^9$ /L. Additionally, patients began 750 mg oral ciprofloxacin twice daily, which was changed to intravenous piperacillin and tazobactam plus liposomal amphotericin B 3.0-5.0 mg/kg/day when the absolute neutrophil count fell below  $0.5 \times 10^9$ /L.

Beginning on the day of hematopoietic stem cell infusion, patients were given subcutaneous granulocyte colony stimulating factor 5 mcg/kg until the absolute neutrophil count was greater than 1.0 x 10<sup>9</sup>/L. For 6 months following transplantation, patients were treated with daily valtrex; fluconazole, voriconazole or itracanozole; and monthly aerosolized pentamidine.

#### Results

Patients transplanted: A total of thirty-one patients, ages 15-53 years, with SLE have undergone transplant. The initial outcomes have been reported in both the New England Journal of Medicine and The Lancet. A report of all 32 patients is in preparation. All were corticosteroid dependent with daily prednisone dose ranging from 60 to 100 mg per day. All had failed between 8 to 18 monthly cycles of IV cyclophosphamide except for patient 2 in whom three cycles of IV cyclophosphamide and plasmapheresis failed to control pulmonary hemorrhage. Post transplant follow-up ranges from 2 to 60 months with a median of 28 months. No patient who underwent HSCT has died. Marked improvement has occurred in organ function for all patients despite gradual withdrawal of all immune suppression. An example of pulmonary improvement post HSCT in all 32 patients follows below.

# DLCO BEFORE AND AFTER HSCT IN 32 SLE PATIENTS UNDERGOING HSCT AT NORTHWESTERN



# 1.5.4. Phase I Study Worldwide

Hematopoietic stem cell transplants for SLE have also been ongoing in Europe. A summary of the European case reports follows in Table 2. These reports have been equally encouraging with remissions up to 3 years.

Table 2: Published Results on HSCT for SLE in Europe

| Disease<br>reference | | Rumber<br>of<br>patients | |
|---|---|---|---|
| SLE (81) | Thiotepa, cyclophosphamide | 1 | Remission for >3 years |
| SLE (82) | Cytoclophosphamide ATG | 2 | Remission for > 12 months |
| SLE (79) | BEAM | 1 | Remission for >1 year |
| SLE (83) | Cyclophosphamide, ATG | 1 | Remission for 8 months |

07-22-2015

# 2. Study Rationale

### 2.1. Selection of Study Population

The phase I study discussed in Section 1.6.3 was designed to select patients with refractory and intractable disease. While those study results were promising, HSCT of patients with impaired visceral organ function and chronic exposure to glucocorticoid therapy is a complicated and high-risk procedure. Enrolling participants earlier in disease who are less ill would also decrease the morbidity and mortality of HSCT. For this reason, the entry criterion for visceral but non-renal involvement is lessened for the current study. Participants with extra-renal lupus need to fail 3 months (instead of 6 months) of monthly cyclophosphamide. For participants in whom the indication is nephritis, active disease must be present despite at least 6 cycles of monthly pulse cyclophosphamide.

# 2.2. Summary of the Known and Potential Risks and Benefits to Human Subjects

#### 2.2.1. Risks

Participation in this trial is associated with certain risks both from the high dose therapy and from the stem cell transplantation.

Cyclophosphamide. The administration of high dose cyclophosphamide is associated with risk of myelosuppression, leukopenia (nadir 8-14 days), hemorrhagic cystitis, syndrome of inappropriate secretion of antidiuretic hormone (SIADH), bladder carcinoma, cellular dysplasias, mucositis, rash, alopecia, anorexia, nausea, vomiting, sterile phlebitis, rare pulmonary toxicity, teratogenicity, hemorrhagic myocarditis, infertility, secondary leukemia; and with rapid IV push oropharyngeal tingling, metallic taste, headache, urticaria, and facial swelling.

Hematopoietic stem cell transplantation: The major hazard of this protocol is transplant-related morbidity and mortality. The marrow suppressive regimen of cyclophosphamide and anti-thymocyte globulin will temporarily destroy the hematopoietic ability of the patient's marrow, and leave the patient susceptible to a wide variety of infections and bleeding complications until the re-infused marrow engrafts. Aggressive supportive care as described above will be used to prevent all avoidable risk. However, a small percentage of participants (expected to be less than 5%, based on previous autologous BMT reported studies) may die as a direct result of transplant related complications. Transplant related mortality is directly related to a participant's age, general medical condition, organ dysfunction, and prior exposure to prolonged or aggressive chemotherapy regimens. Transplant related complications include infections, bleeding, veno-occlusive disease of the liver, and failure to engraft.

<u>Risk from rabbit ATG/rituximab</u>: "serum sickness" (a hypersensitivity reaction consisting of fever, rashes, joint pain and kidney disease); anaphylaxis

(sudden and severe allergic reaction that could result in death); chills, pains in your joints, headache, muscle pain, nausea, vomiting, diarrhea, chest-pain, low blood pressure, shortness of breath, fluid in the lungs, abdominal pain; abnormal liver function and renal function; and low blood platelet count. Low CD4+ counts may also occur and may result in death related to infection.

Risk from G-CSF: myalgias, headache, flu-like symptoms, fever, bone pain in approximately 20% of participants, possible elevation of uric acid, transaminases, and LDH.

Risk from Leukapheresis: This procedure requires 4-6 hours and will be performed through the pheresis catheter or a 16-gauge catheter introduced into the antecubital vein. The total volume outside the body at any time does not exceed 450 ml. The most common complication is hypocalcemia arising from citrate anticoagulation, which is usually mild or rarely severe with nausea, vomiting or arrhythmias. Symptoms are avoided with replacement solutions added during apheresis, slowing the flow rate, and/or supplemental oral antacids containing calcium. Other complications are infrequent, but include hypotension, vasovagal syncope and infection.

<u>Central Line</u>: Placement of an external central line catheter device is a routine procedure, which may be done under local or general anesthesia. Potential complications include bleeding, pneumothorax, hemothorax, or arrhythmia. Like all artificial devices, lines may become infected and require treatment with antibiotics and/or removal.

#### 2.2.2. Benefits

If the phase I results can be replicated, participants who receive SCT should benefit with corticosteroid-free remissions for three or more years. This is in contrast to participants who receive treatment with cyclophosphamide, many of whom will continue to have active disease requiring treatment.

### 3. Objectives

This trial is designed to evaluate the safety of treating systemic lupus erythematosus participants with high dose cyclophosphamide and rATG/rituximab immune ablation, followed by rescue with unmanipulated peripheral stem cells.

# 4. Endpoints and Outcomes

# 4.1. Primary Outcome

The primary efficacy outcome is overall survival and the proportion of participants who achieve and maintain remission after transplant. Remission is defined according to the RIFLE as duration on no immune suppressive medications except physiologic doses of prednisone (<10 mg/day) or corticosteroid equivalent and or hydroxychloroquine

### 4.2. Secondary Outcomes

The secondary efficacy outcomes include the following:

- 1) Serology, ANA titer, anti-ds DNA antibody titer, and C3 and C4
- 2) SLEDAI
- 3) CrCl and DLCO Adj

# 5. Study Design and Populations

### 5.1 Study Population

Participants meeting the inclusion and exclusion criteria specified below may be enrolled.

#### 5.1.1. Inclusion Criteria

The inclusion criteria are:

- Ages 15 to 60 years old
- Meet at least 4 of 11 American College of Rheumatology (ACR)
   Classification criteria for SLE (see Appendix 16.2)
- Meet one of following five:
  - a) For lupus nephritis, participants must fail pulse cyclophosphamide (500 to 1000 mg/m² monthly for a minimum of 6 months) or cell cept. Failure is defined as meeting criteria to be considered as BILAG renal category A.
  - b) For visceral organ involvement other than nephritis, participants must be BILAG cardiovascular/respiratory category A, vasculitis category A, or neurologic category A and must fail at least 3 months of oral or IV cyclophosphamide and be corticosteroid dependent. Steroid dependence being defined as at least 3 months of steroid therapy and inability to wean corticosteroid to less than 20 mg/day of prednisone or equivalent.

- c) For cytopenias that are immune mediated, participants must be BILAG hematologic category A. Participants must fail corticosteroids (either oral prednisone > 0.5 mg/kg/day for more than 6 months or pulse methylprednisolone for at least one cycle of three days), and at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, mycophenolate mofetil 2 grams daily for more than 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months, danazol for at least 3 months, or splenectomy.
- d) For mucocutaneous disease, participants must meet BILAG mucocutaneous category A, be unable to be weaned from prednisone to less than 0.5 mg/kg/day for more than 6 months and obvious Cushingoid habitus, and have received at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, methotrexate at 15mg/week for at least 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months.
- e) For arthritis/myositis, participants must meet BILAG musculoskeletal category A, be unable to be weaned from prednisone to less than 0.5 mg/kg/day for more than 6 months and obvious Cushingoid habitus, and have received at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, methotrexate at 15mg/ week for at least 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months.
- Able to give informed consent.
- If indication for HSCT is nephritis, a renal biopsy must demonstrate the
  potential of a reversible (non-fibrotic) component indicating that if
  successful the participant would not be likely to be permanently dialysisdependent after transplant.
- Since the BILAG is only one of multiple indices for SLE, patients may also be candidates if despite prior immune suppression therapy as described above, patients are still on active immune suppression (more than 10mg a day of prednisone).
- Patients with SLE whose major manifestation is Antiphospholipid syndrome (APS) may be candidates without prior immune suppression therapy if they have had a visceral organ thrombotic or embolic event despite anticoagulation.

# 5.1.2. Exclusion Criteria

- HIV positive
- Ongoing malignancy except localized basal cell or squamous skin cancer.
   Other malignancies for which the participant is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I or II breast

cancer will be considered on an individual basis by the investigators doing the final screening for participant qualification.

- Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
- Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
- DLCO < 45% of predicted unless attributed to active lupus.
- Resting LVEF < 40% unless attributed to active lupus.</li>
- Known hypersensitivity to E Coli derived proteins.
- Transaminases greater than 2 times normal unless attributed to active lupus.
- Positive tuberculosis skin test
- Anv active infection
- Any co-morbid illness that in the opinion of the investigator would jeopardize the ability of the subject to tolerate the study.
- Failure to collect at least 2.0 x 10<sup>8</sup> CD34+ cells/kg
- ANA-negative

# 6. Study Treatment and Concomitant Therapies

#### 6.1. Preparation, Administration and Dosage of Study Treatment

#### 6.1.1. Mobilization

Participants will be administered Cyclophosphamide at 2.0 g/m² in 200 ml of normal saline (NS) over 1 hour. Hydration with 0.9 NS at approximately 100-250-ml/ hour will begin 4 hours prior to cyclophosphamide and continued for 24 hours after termination of cyclophosphamide. Urine output approximately greater than 100 ml/hour should be maintained.

G-CSF will be administered subcutaneously at 5-10 mcg/kg/day and will be started 5 days after termination of cyclophosphamide administration.

After the absolute neutrophil count is greater than 1000/ul or after hematological nadir, leukapheresis using a continuous flow blood cell separator will be initiated. A 10-15 liter apheresis will be performed unless stopped earlier for clinical judgment of toxicity (e.g., numbness, tetany). The G-CSF will continue until apheresis is discontinued. If necessary, platelets will be transfused to greater than 60,000/ul prior to each apheresis.

Table 3: Stem Cell Mobilization with Cyclophosphamide and G-CSF

| DAY | 0 | 1 | 2 | 3 | 4 | 5 | 10 | ANC >1.0 |
|--------------------------------------|---|---|---|---|---|---|----|----------|
| Cyclophosphamide 2 gm/m <sup>2</sup> | X | | | | | | | |
| G-CSF<br>(5-10 mcg/kg/day) | | | | X | Х | X | X | X |
| Apheresis* | | | | | | | | X |

<sup>\*</sup> Apheresis begins when ANC >  $1.0 \times 10^9$ /L and continues until >2.0 x  $10^6$  CD34 cells/kg patient weight are cryopreserved. A maximum of 4 apheresis may be performed. If the minimum number of CD34 cells ( $2.0 \times 10^6$  /kg) have not been collected, the patient will not receive the conditioning regimen or HSCT.

# 6.1.2. Conditioning Regimen

**Table 4. Conditioning Regimen** 

| Day | -6 | -5 | -4 | -3 | -2 | -1 | 0 | +1 | +6 |
|---|---|---|---|---|---|---|---|---|---|
| Hydration | X | X | X | X | X | | T | | |
| Cyclophosphamide (50 mg/kg/d) | | Х | X | Х | Х | | | | |
| Mesna | | X | X | Х | X | | | | |
| Rabbit ATG<br>(mg/kg/d) IV | | 0.5 | 1 | 1.5 | 1.5 | 1.5 | | | |
| Solumedrol 250 mg | | Х | Х | Х | Х | Х | | | |
| Rituximab 500mg/d<br>IV | X | | | | | | | Х | |
| Stem Cells infused | | | | | | | X | | |
| G-CSF<br>5mcg/kg/d start D+6 | | | | | | | | | Х |

<u>Hydration</u>: approximately 50-200cc/hour in adults should begin 6 hours before cyclophosphamide and continue until 24 hours after the last cyclophosphamide dose. Hydration rates need to be individually adjusted by daily weights to maintain dry weight count. BID weights will be obtained. **Warning:** Participants with renal insufficiency are prone to volume overload. Early institution of ultrafiltration or dialysis is recommended.

Cyclophosphamide: 50 mg/kg/day x 4 days (the lesser of ideal or actual weight) will be given intravenously over 1 hour in 250 cc of normal saline on days -5 through -2.

Mesna: 50mg/kg/day x 4 days will be given intravenously over 24 hours.

Rabbit ATG 0.5mg/kg will be given IV on day -5, 1.0mg/kg will be given on day -4, 1.5mg/kg will be given IV on days -3, -2, -1 (no dose adjustment). It will be given over 10 hours. Premedicate with Solumedrol 250mg IV, acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion.

Rituximab 500mg/day will be given IV on days –6 and +1. At the first dose (D-6), rituximab infusion will be started at 50mg/h and escalate the infusion rate by 50mg every 30minutes to a maximum of 400mg/h. Starting the second dose (days –4, -2 and +1). IV infusion will be started at 100mg/h and escalate the infusion rate 100mg every 30minutes to a maximum of 400mg/h. Premedicate with Solumedrol 250mg IV, acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion on days –6 and +1. Premedicate acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion on days –4 and –2.

<u>G-CSF</u> will be continued until absolute neutrophil count reaches at least 1,000cells/ml for three days

#### 6.1.3. Stem Cell Reinfusion

Previously collected stem cells will be reinfused on day 0 as noted in Table 4. The stem cells are infused over approximately 20 minutes through the central venous catheter (e.g., PICC line). Following stem cell reinfusion, routine daily labs will be obtained including CBC, chemistry panel, and liver function tests. Antibiotics and blood transfusions will be administered as required by clinical judgment.

#### 6.1.4. Infection Prophylaxis Guidelines

All prophylactic antibiotics may be changed or discontinued according to clinical circumstances (such as patient allergy) as determined by attending physician(s).

Antibacterial prophylaxis - Ciprofloxacin 500 mg po BID from day -10 until neutrophil count is less than 500/ul. When ANC is < 500/ul, a broad-spectrum intravenous antibiotic such as Zosyn or Cefepime is recommended regardless of temperature until ANC returns to > 500/ul. Aerosolized pentamidine 300mg will be given monthly for 6 months (bacterial and pneumocystis prophylaxis).

<u>Antifungal prophylaxis</u> – Either Voriconazole 200 mg bid or Ambisome 5mg/kg will be given while neutropenic during both mobilization and transplantation. When

ANC is > 500/ul, Voriconazole is recommended for a minimum of 6 months or longer until the participant is tapered off corticosteroids.

Antiviral prophylaxis – Valtrex 500 mg po TID from day of admission until ANC > 500/ul. Oral valganciclovir (dose adjusted for Cr, WBC and platelets) will be given until day 90. Thereafter, Valtrex is recommended for a minimum of one year or longer until the participant is tapered off corticosteroids.

#### 6.1.5. Transfusion Guidelines

Since SLE may have a vasculitis component, the platelet count should be maintained over 30,000/ul throughout the transplant period.

# 6.2. Modification and Discontinuation of Study Treatment or Study Protocol Procedures

All prophylactic antibiotics indicated in Section 6.1.2 may be changed or discontinued according to clinical circumstances (such as patient allergy) as determined by attending physician(s).

The investigator must apply his/her clinical judgment to determine if an adverse event is of sufficient severity to require that the subject should immediately be removed from treatment. If necessary, an investigator must suspend any trial treatments and institute the necessary medical therapy to protect a subject from any immediate dangers.

# 7.0 Study Parameters—all pre-transplant tests must be obtained within 3 months of study entry

| Test / evaluation | Pre-<br>enrollment | Upon<br>admission<br>for HSCT | During<br>hospitaliz<br>ation | Weekly for 4<br>weeks after<br>transplant | 6 mo, 12 mo,<br>then yearly for 5<br>years* |
|---|---|---|---|---|---|
| History and physical | Х | X | DAILY<br>SOAP | X | Х |
| Medications /dose | X | X | X | Х | X |
| SLEDAI | X | | | | X |
| CXR, EKG | X | | | | X (if clinically indicated) |
| CBC with diff | X | X | X daily | X | X |
| Electrolytes and Cr | X | X | X daily | X | X |
| AST, ALT, bili, alk phos | Х | Х | X three<br>times a week | Х | Х |
| Dobutamine stress Doppler echocardiography | X | | | | X (dobutamine optional) |
| ANA, anti-ds DNA, Anti-<br>SSA, SSB, anti-Sm | X | | | | X |
| ACLA IGG, IGM, Anti-<br>beta-2 glycoprotein, LA | X | | | | Х |
| C3, C4 | X | | | | X |
| PT, PTT | X | | | | |
| Hepatitis A, B, C, HTLV-<br>I, HTVL-III, CMV titer | X | | | | |
| UA, 24 hour urine CrCl and protein | Х | | | | X(if clinically indicated) |
| PFT with DLCO | X | | | | X |
| HRCT | X (only if clinically indicated) | | | | X (only if clinically indicated) |
| Marrow biopsy and aspirate (as indicated for patients with cytopenias | X | | | | X (only if clinically indicated) |
| Pregnancy test | X | X | | | |
| Dental consultation | X | | | | |
| CT scan of sinuses | X (optional) | | | | |
| Neurocognitive | X (only if indicated for active cerebritis) | | | | X (only if indicated for active cerebritis) |
| MRI with gad and/or<br>MRA of brain | X (if indicated for active cerebritis) | | | | X (only if clinically indicated) |
| Quality of life scale (SF-36) | X | | | | X |

<sup>\*</sup> EVERY EFFORT WILL BE MADE TO HAVE THE PATIENT RETURN FOR FOLLOW-UP, HOWEVER, IF PATIENT CANNOT RETURN FOR FOLLOW-UP, STUDY TESTS AND MEDICAL EVALUATION WILL BE COLLECTED FROM LOCAL PHYSICIAN AS WELL AS TELEPHONE HISTORY BY STUDY PHYSICIAN AND PROTOCOL NURSE.


#### 7.1 HOSPITAL DISCHARGE GUIDELINES

- 1) Afebrile with no evidence of active infection
- 2) Transfusion independent or requiring less than one platelet and or PRBC transfusion per week
- 3) Adequate oral nutrition
- 4) Complies with outpatient follow-up schedule, visiting nurse (if required), and labs

#### 8.0 EVALUATION OF TOXICITY

Assessment will be made with regards to toxicity by one of the protocol investigators. Common Toxicity Criteria Scale (see appendix) will be used to grade all non-hematologic toxicities.

### 9.0 ADVERSE EVENT REPORTING

The Toxicity grading for adverse events is according to NCI common toxicity criteria for adverse events (CTCAE) version 2.0 at website http://ctep.info.nih.gov (besides being located on the website, CTC v2.0 providing an alphabetical listing of Adverse Events with associated descriptions to grade severity is attached at end of the protocol)

- 9.1 <u>To be reported by phone (312-695-4960) or FAX (312-695-4961) to</u> Richard Burt:
  - a) All life-threatening or lethal (Grade 4 and 5) (except grade 4 myelosuppression which is anticipated) reactions. This information is to be immediately reported to Dr Richard Burt who will report it within 72 hours of a working day to the IRB and FDA.
- 9.2 <u>To be reported in writing within 10 working days to Richard K</u> Burt (312-695-4960)
  - a) Grade 3 reactions. These will be reported by Dr. Burt on annual reports to the FDA.

# 10.0 Follow-up procedures for withdrawal subjects

Unless the patient refuses, subjects who withdraw from the study will be followed in a manner consistent with the monitoring plan.

### 11.0 Statistical Considerations

This is a phase II study of 40 patients. Statistical considerations and safety rules for the protocol are as follows:

- 11.1 Stopping rules for transplant-related regimen-related toxicity.

  Regimen-related toxicity within the first 28 days after transplant will be determined as follows: non-hematological grade 4 toxicity that fails to resolve in 10 days; and hematological grade 4 toxicity that fails to resolve in 28 days. Operationally sufficient evidence of any ratio of regimen-related toxicity will occur when any of the following ratios is observed: any 2/6 or 4/10, or 6/40.
- 11.2 Stopping rules for transplant-related mortality (TRM). TRM will be defined as death within the first 100 days of transplant due to transplant-related complications. Operationally, this will occur with any 2 of 10 deaths, or 4/40.
- 11.3 Any death within the first 100 days will result in halting the study until reviewed and the IRB and FDA notified.

#### 12.0 Literature References

- Rus V and Hochberg MC, The epidemiology of SLE. In Dubois' Lupus Erythematosus, 6<sup>th</sup> ed. Edited by Wallace D and Hahn BH, Lippincott, William and Wilkens, Philadelphia, 2002 in press.
- Urowitz MB, Gladman DD, Abu-Shakra M et al. Mortality studies in SLE. Results from a single center. III. Improved survival over 24 years. J Rheumatol 1997; 24:1061-5.
- 3. Rose NR. and Bona C. Defining criteria for autoimmune diseases (Witebsky's postulates revisited) *Immunology Today* 1993; 14(9):426-429.
- Dang H, Harbeck RJ. The in vivo and in vitro glomerular deposition of isolated anti-double-stranded DNA antibodies in NZB/W mice. Clin Immunol Immunopathol 1984; 31: 265-278.
- Tsao, B., Kronenberg, M., Cheroutre, H., and Hahn, B.H. Failed self-tolerance and autoimmunity in mice transgenic for an IgG anti-DNA. J. Immunol. <u>149</u>:350-358, 1992.
- 6. Ehrenstein MR, Katz DR, Griffiths M, Winkler TH, Kalden JR, Isenberg DA. Human monoclonal IgG anti-DNA antibodies deposit in kidneys and induce proteinuria in SCID mice (abst). *Lupus* 1995; 4 (Suppl 2): 69.
- 7. Marmont AM. The transfusion of active LE plasma into nonlupus recipients, with a note on the LE-like cell. *Annals New York Academy of Sciences*, 1965; 124(2): 838-851.
- 8. Ward MM, Pisetsky DS, Christenson VD. Antidouble stranded DNA antibody assays in systemic lupus erythematosus: correlations of longtitudinal antibody measurements. *J Rheumatol* 1989; 16: 609-613.
- Symmons DPM, Coopock JS, Bacon PA, Bresnihan B, Isenberg DA, Maddison P, Mchugh N, Snaith ML, Zoma AS. Development and assessment of a computerized index of clinical disease activity in systemic lupus erythematosus. QJ Med 1988; 68: 927-937.
- Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The committee on prognosis studies in SLE. Arthritis Rheum 1992; 35: 630-640.
- 11. Liang MH, Socher SA, Roberts WN, Esdaile JM. Measurement of systemic lupus erythematosus activity in clinical research. *Arthritis Rheum* 1988; 31: 817-825.
- Petri M, Bochemstedt L, Colman J, Whiting-O'Keefe Q, Fitz G, Sebastin A, Hellman D. Serial assessment of glomerular filtration rate in lupus nephropathy. Kidney Int 1988; 34: 832-839
- 13. Gladman DD, Goldsmith, C.H, Urowitz MB, Bacon, P.A, Bombardier C, Isenberg, D, Kalunian K, Liang, MH, Maddison, P, Nived, O, Richter, M, Snaith, M, Symmons, D, Zoma, A. Cross-cultural validation and reliability of three disease activity indices in systemic lupus erythematosus. *J Rheum* 19:608-611, 1992.
- 14. Gladman DD, Goldsmith CH, Urowitz MB, Bacon PA, Bombardier C, Isenberg D, Kalunian K, Liang MH, Maddison P, Nived O, Richter M, Snaith M, Symmons D, Zoma A. Sensitivity to change of three SLE disease activity indices: international validation. *J Rheum* 21:14568-1471, 1994.

- 15. Watson ML. Rao JK. Gilkeson GS. Ruiz P. Eicher EM. Pisetsky DS. Matsuzawa A. Rochelle JM. Seldin MF. Genetic analysis of MRL-lpr mice: relationship of the Fas apoptosis gene to disease manifestations and renal disease-modifying loci. *Journal of Experimental Medicine*. 1992; 176(6):1645-56.
- 16. Vidal S. Kono DH. Theofilopoulos AN. Loci predisposing to autoimmunity in MRL-Fas lpr and C57BL/6-Faslpr mice. *Journal of Clinical Investigation*. 1998; 101(3):696-702.
- Drake CG. Babcock SK. Palmer E. Kotzin BL. Genetic analysis of the NZB contribution to lupus-like autoimmune disease in (NZB x NZW) F1 mice.
   Proceedings of the National Academy of Sciences of the United States of America. 1994; 91(9):4062-6.
- 18. Morel L. Mohan C. Yu Y. Croker BP. Tian N. Deng A. Wakeland EK. Functional dissection of systemic lupus erythematosus using congenic mouse strains. Journal of Immunology. 158(12):6019-28, 1997 Jun 15.
- Kono DH. Burlingame RW. Owens DG. Kuramochi A. Balderas RS. Balomenos D. Theofilopoulos AN. Lupus susceptibility loci in New Zealand mice. Proceedings of the National Academy of Sciences of the United States of America. 91(21):10168-72, 1994 Oct 11.
- 20. Mohan C. Morel L. Yang P. Wakeland EK. Genetic dissection of systemic lupus erythematosus pathogenesis: Sle2 on murine chromosome 4 leads to B cell hyperactivity. Journal of immunology. 159(1):454-65, 1997 Jul 1
- 21. Mohan C. Alas E. Morel L. Yang P. Wakeland EK. Genetic dissection of SLE pathogenesis. Sle1 on murine chromosome 1 leads to a selective loss of tolerance to H2A/H2B/DNA subnucleosomes. Journal of Clinical Investigation. 101(6):1362-72, 1998 Mar 15.
- 22. Autoantibody-inducing T helper lines from patients with active lupus nephritis: isolation of CD8-T helper cell lines that express the gamma delta T-cell antigen receptor. *Proc Natl Acad Sci* USA 1990; 87: 7020.
- 23. Tsao BP and Hahn BH. Systemic lupus erythematosus. In *Emery and Rimoin's Principles and practice of Medical Genetics*, 4<sup>th</sup> Edition. 2001. In press.
- 24. Dubois EL, Commons RR, Star P, Stein CS Jr, Morrison R. Corticotropin and cortisone treatment for systemic lupus erythematosus. *JAMA* 1952; 149: 995-1002.
- 25. The epidemiology of SLE. In Dubois' Lupus Erythematosus, 5th ed. Edited by Wallace D and Hahn BH, Williams and Wilkens, Baltimore, 1997, pp49-68.
- 26. Traynor AE. Schroeder J. Rosa RM. Cheng D. Stefka J. Mujais S. Baker S. Burt RK. Treatment of severe systemic lupus erythematosus with high-dose chemotherapy and haemopoletic stem-cell transplantation: a phase I study. Lancet. 356:701-7, 2000
- 27. Vassilopoulos D, Kovacs B, Tsokos GC. TCR/CD3 complex-mediated signal transduction pathway in T cells and cell lines from patients with systemic lupus erythematosus. *J Immunol* 1995; 155: 2269.
- 28. Liossis SN, Ding DZ, Dennis GJ, Tsokos GC. Altered pattern of TCR/CD3-mediated protein-tyrosyl phosphorylation in T cells from patients with systemic lupus erythematosus. Deficicent expression of the T cell receptor zeta chain. *J Clin Invest* 1998; 101: 1448.

- 29. Rengaraju M, Gray JD, Horwitz DA, Kubin M, Trinchierir G. Increased spontaneous IL-10 production and decreased mitogen-induced INF□ and TNF□ production in untreated patients with SLE; role of CD8+ T cells. Lupus 1995; 4(suppl2): 82.
- 30. Koshy M, Berger D, Crow MK. Increased expression of CD40L on Sie lymphocytesa, J Clin Invest 1996;95:526-37.
- 31. Vakkalanka RK, Woo C, Kirou KA, Berger D, Crow M. Elevated levels and functional capacity of soluble CD40L in SLE sera. Arthritis Rheum 1999; 42:871-8.
- 32. Grennan DM. Parfitt A. Manolios N. Huang Q. Hyland V. Dunckley H. Doran T. Gatenby P. Badcock C. Family and twin studies in systemic lupus erythematosus. Disease Markers. 13(2):93-8, 1997 Apr.
- 33. Horwitz DA, Stohl W and Gray JD. T lymphocytes, natural killer cells, cytokines and immune regulation in Dubois' Lupus Erythematosus 5<sup>th</sup> ed. Edited by Wallace D and Hahn BH, Williams and Wilkens, Baltimore, 1997, pp 155-194: updated 6<sup>th</sup> edition in press.
- 34. Cross JT; Benton HP. The roles of interleukin-6 and interleukin-10 in B cell hyperactivity in systemic lupus erythematosus. (Inflammation Research, 1999 May, 48(5):255-61).
- 35. Traynor AE, Schroeder J, Rosa RM, Cheng D, Stefka J, Mujais S, Baker S, Burt RK. Treatment of severe systemic lupus erythematosus with high-dose chemotherapy and haemopoietic stem cell transplantation. A phase I study. [comment]. *Lancet*. 356(9231): 701-7, 2000 Aug 26.
- 36. Traynor AE, Barr WG, Rosa RM, Rodriguez J, Oyama Y, Baker S, Brush M, Burt RK. Hematopoietic stem cell transplantation for severe and refractory lupus. Analysis after five years and fifteen patients. *Arthritis and Rheumatism.* 46(11): 2917-23, 2002.
- Ben-Asher S. Recurrent acute lupus erythematosus disseminatus: report of case, which has survived 23 years after onset of systemic manifestations. *Ann Intern Med* 1951; 34: 243-248.
- 38. Wallace DJ, Podell T, Weiner J, Klinenberg JR, Forouzesh S, Duboius EL. Systemic lupus erythematosus-survival patterns. Experience with 609 patients. *JAMA* 1981 6; 245: 934-938.
- 39. Steinberg AD, Stenberg SC. Long-term preservation of renal function in patients with lupus nephritis receiving treatment that included cyclophosphamide versus those treated with prednisone only. *Arthritis Rheum* 1991; 34:945-50.
- 40. Chan TM; Li FK; Tang CS; Wong RW; Fang GX; Ji YL; Lau CS; Wong AK; Tong MK; Chan KW; et al. Efficacy of mycophenolate mofetil in patients with diffuse proliferative lupus nephritis. Hong Kong-Guangzhou Nephrology Study Group. New Eng J Med, 2000; 343(16):1156-62.
- 41. Burt RK. Padilla J. Dal Canto MC. Miller SD. Viral hyperinfection of the central nervous system and high mortality after hematopoietic stem cell transplantation for treatment of Theiler's murine encephalomyelitis virus-induced demyelinating disease. *Blood.* 1999; 94(8):2915-22.
- 42. Van Bekkum DW. Stem cell transplantation in experimental models of autoimmune disease. *Journal of Clinical Immunology*. 2000; 20(1):10-6.

- 43. Karussis D. Vourka-Karussis U. Mizrachi-Koll R. Abramsky O. Acute/relapsing experimental autoimmune encephalomyelitis: induction of long lasting, antigenspecific tolerance by syngeneic bone marrow transplantation. *Multiple Scierosis*. 1999; 5(1):17-21.
- 44. Kamiya M. Sohen S. Yamane T. Tanaka S. Effective treatment of mice with type II collagen induced arthritis with lethal irradiation and bone marrow transplantation. *Journal of Rheumatology*. 1993; 20(2):225-30.
- 45. Burt RK. Padilla J. Begolka WS. Canto MCD. Miller SD. Effect of disease stage on clinical outcome after syngeneic bone marrow transplantation for relapsing experimental autoimmune encephalomyelitis. *Blood.* 1998; 91(7):2609-16.
- 46. van Gelder M. van Bekkum DW. Effective treatment of relapsing experimental autoimmune encephalomyelitis with pseudoautologous bone marrow transplantation. *Bone Marrow Transplantation*. 1996; 18(6):1029-34.
- 47. Blank M. Tomer Y. Slavin S. Shoenfeld Y. Induction of tolerance to experimental anti-phospholipid syndrome (APS) by syngeneic bone marrow cell transplantation. *Scandinavian Journal of Immunology*. 1995; 42(2):226-34.
- 48. Karussis DM. Vourka-Karussis U. Lehmann D. Abramsky O. Ben-Nun A. Slavin S. Immunomodulation of autoimmunity in MRL/lpr mice with syngeneic bone marrow transplantation (SBMT). *Clinical & Experimental Immunology*. 1995;100(1):111-7.
- 49. Karussis DM. Vourka-Karussis U. Lehmann D. Ovadia H. Mizrachi-Koll R. Ben-Nun A. Abramsky O. Slavin S. Prevention and reversal of adoptively transferred, chronic relapsing experimental autoimmune encephalomyelitis with a single high dose cytoreductive treatment followed by syngeneic bone marrow transplantation. *Journal of Clinical Investigation*. 1993; 92(2):765-72.
- 50. van Gelder M. Kinwel-Bohre EP. van Bekkum DW. Treatment of experimental allergic encephalomyelitis in rats with total body irradiation and syngeneic BMT. *Bone Marrow Transplantation*. 1993; 11(3):233-41.
- 51. Van Bekkum DW. BMT in experimental autoimmune diseases. *Bone Marrow Transplantation*. 1993; 11(3):183-7.
- 52. Pestronk A. Drachman DB. Teoh R. Adams RN. Combined short-term immunotherapy for experimental autoimmune myasthenia gravis. *Annals of Neurology*. 1983; 14(2):235-41.
- 53. Kirzner RP; Engelman RW; Mizutani H; Specter S; Good RA. Prevention of coronary vascular disease by transplantation of T-cell-depleted bone marrow and hematopoietic stem cell preparation in autoimmune-prone w/BF (1) mice. Biology of Blood and Marrow Transplantation. 2000; 6(5):513-22.
- 54. Wang B; Yamamoto Y; El-Badri NS; Good RA. Effective treatment of autoimmune disease and progressive renal disease by mixed bone-marrow transplantation that establishes a stable mixed chimerism in BXSB recipient mice. *Proc Natl Acad Sciences USA*, 1999 Mar 16, 96(6):3012-6.
- 55. Bielschowsky M, Helyer BJ, Howie JB. Spontaneous haemolytic anaemia in mice of the NZB/BI strain. *Proc Univ Otago Med Sch* (NZ) 1959; 37: 9-11.
- 56. Yoshida S, Castles JJ, Gershwin ME. The pathogenesis of autoimmunity in New Zealand mice. Semin Arthritis Rheum 1990; 19: 224-242.

- 57. Kono DH, Burlingame RW, Owens DG, Kuramochi A, Balderas RS, Balomenos D, Theofilopoulos AN. Lupus susceptibility loci in New Zealand mice. *Proc Natl Acad Sci USA* 1994; 91:10168-10172.
- 58. Eastcott JW, Scxhwartz RS, Datta SK. Genetic analysis of the inheitance of B cell hyperactivity in relation to the development of autoantibodies and glomerulonephritis in NZB x SWR crosses. *J Immunol* 1983; 131: 2232-2239.
- 59. Murphy ED, Roths JB. A single gene for massive lymphoproliferation with immune complex disease in a new mouse strain MRL. In: Proceedings of the 16th International Congress in Hematology. Amsterda: Excerpta Medica, 1976: 69-80.
- 60. Watanabe-Fukunaga R, Brannan CI, Copeland NG, Jenkins NA, Nagata S. Lymphoproliferative disorder in mice explained by defects in Fas antigen that mediates apoptosis. *Nature* 1992; 356: 314-317.
- 61. Makin M, Fumiwara M, Watanabe H. Studies on the mechanisms of the development of lupus nephritis in BXSB mice. I. Analysis of immunological abnormalities at the onset period. *J Clin Lab Immunol* 1987; 22: 127-131.
- 62. Murphy ED, Roths JB. A Y chromosome associated factor in strain BXSB producing accelerated autoimmunity and lymphoproliferation. *Arthritis Rheum* 1979; 22: 1188-1194.
- 63. Hashimoto Y, Kawamura M, Ichikawa K, Suzuki T, Sumida T, Toshida S, Matsuura E, Ikehara S, Koike T. Anticardiolipin antibodies in NZW x BXSB F1 mice. A model of antiphospholipid syndrome. *J Immunol* 1992; 149: 1063-1068.
- 64. Ikehara S, Nakamura T, Sekita K, Muso E, Hasunizu R, Ohtsuki H, Hamashima Y, Good R, treatment of systemic and organ-specific autoimmune disease in mice by allogeneic bone marrow transplantation. *Prog Clin Biol Res* 1987; 229: 131-146.
- 65. Himeno K, Good RA. Marrow transplantation from tolerant donors to treat and prevent autoimmune diseases in BXSB mice. *Proc Natl Acad Sci USA* 1988; 85: 2235-2239.
- 66. Karussis DM, Vourka-Karussis U, Lehmann D, Abramsky O, Ben-Nun A, Slavin S. Immunomodulation of autoimmunity in MRL/lpr mice with syngeneic bone marrow transplantation (SBMT). *Clin Exp Immunol* 1995; 100:111-117.
- 67. Ishida T, Inaba M, Hisha H, Sugiura K, Adachi Y, Nagata N, Ogawa R, Good RA, Ikahara S. Requirement of donor-derived stromal cells in the bone marrow for successful allogeneic bone marrow transplantation. Complete prevention of recurrence of autoimmune diseases in MRL/MP-Ipr/Ipr mice by transplantation of bone marrow plus bones (stromal cells) from the same donor. *J Immunol* 1994; 152: 3119-3127.
- 68. Demirer T. Celebi H. Arat M. Ustun C. Demirer S. Dilek I. Ozcan M. Ilhan O. Akan H. Gurman G. Koc H. Autoimmune thrombocytopenia in a patient with small cell lung cancer developing after chemotherapy and resolving following autologous peripheral blood stem cell transplantation. Bone Marrow Transplantation. 1999; 24(3):335-7.
- 69. Jindra P. Koza V. Fiser J. Vozobulova V. Svojgrova M. Autologous CD34+ cells transplantation after FAMP treatment in a patient with CLL and persisting AIHA:

- complete remission of lymphoma with control of autoimmune complications. Bone Marrow Transplantation. 1999; 24(2):215-7.
- 70. Schachna L. Ryan PF. Schwarer AP. Malignancy-associated remission of systemic lupus erythematosus maintained by autologous peripheral blood stem cell transplantation. *Arthritis & Rheumatism*, 1998; 41(12):2271-2.
- 71. Rosler W. Manger B. Repp R. Kalden JR. Gramatzki M. Autologous PBPCT in a patient with lymphoma and Sjogren's syndrome: complete remission of lymphoma without control of the autoimmune disease. *Bone Marrow Transplantation*. 1998; 22(2):211-3.
- 72. Skoda RC. Tichelli A. Tyndall A. Hoffmann T. Gillessen S. Gratwohl A. Autologous peripheral blood stem cell transplantation in a patient with chronic autoimmune thrombocytopenia. *British Journal of Haematology*. 1997; 99(1):56-7.
- 73. Cooley HM. Snowden JA. Grigg AP. Wicks IP. Outcome of rheumatoid arthritis and psoriasis following autologous stem cell transplantation for hematologic malignancy. *Arthritis & Rheumatism.* 1997; 40(9):1712-5.
- 74. Snowden JA. Patton WN. O'Donnell JL. Hannah EE. Hart DN. Prolonged remission of longstanding systemic lupus erythematosus after autologous bone marrow transplant for non-Hodgkin's lymphoma. *Bone Marrow Transplantation*. 1997; 19(12):1247-50.
- 75. Meloni G. Capria S. Vignetti M. Mandelli F. Modena V. Blast crisis of chronic myelogenous leukemia in long-lasting systemic lupus erythematosus: regression of both diseases after autologous bone marrow transplantation. *Blood.* 1997; 89(12):4659.
- 76. Euler HH. Marmont AM. Bacigalupo A. Fastenrath S. Dreger P. Hoffknecht M. Zander AR. Schalke B. Hahn U. Haas R. Schmitz N. Early recurrence or persistence of autoimmune diseases after unmanipulated autologous stem cell transplantation. *Blood.* 1996; 88(9):3621-5.
- 77. De Stefano P. Zecca M. Giorgiani G. Perotti C. Giraldi E. Locatelli F. Resolution of immune haemolytic anaemia with allogeneic bone marrow transplantation after an unsuccessful autograft. *British Journal of Haematology*. 1999; 106(4):1063-4.
- 78. Burt RK. Traynor AE. Pope R. Schroeder J. Cohen B. Karlin KH. Lobeck L. Goolsby C. Rowlings P. Davis FA. Stefoski D. Terry C. Keever-Taylor C. Rosen S. Vesole D. Fishman M. Brush M. Mujias S. Villa M. Burns WH. Treatment of autoimmune disease by intense immunosuppressive conditioning and autologous hematopoietic stem cell transplantation. *Blood*. 1998; 92(10):3505-14.
- 79. Fouillard L, Gorin NC, Laporte JP, Leon A, Brantus JF, Miossec P. Control of severe systemic lupus erythematosus after high-dose immunosuppressive therapy and transplantation of CD34+ purified autologous stem cells from peripheral blood. *Lupus*. 1999; 8(4):320-3.
- 80. Burt RK, Traynor A, Ramsey-Goldman R. Hematopoietic stem-cell transplantation for systemic lupus erythematosus. *N Engl J Med.* 1997 Dec 11; 337(24):1777-8.
- 81. Marmont AM, van Lint MT, Gualandi F, Bacigalupo A. Autologous marrow stem cell transplantation for severe systemic lupus erythematosus of long duration. *Lupus*. 1997; 6(6):545-8.

- 82. Rosen O, Theil A, Massenkeil G, et. al. Autologous stem cell transplantation in refractory autoimmune diseases after ex vivo depletion of mononuclear cells. *Arthritis Res* 2000; 2: 327-336.
- 83. Musso M, Porretto F, Crescimanno A, Bondi F, Polizzi V, Scalone R, Mariani G. Autologous peripheral blood stem and progenitor (CD34+) cell transplantation for systemic lupus erythematosus complicated by Evans syndrome. *Lupus.* 1998; 7(7):492-4.

# 13.0 Appendices

DI SLE.Auto2003

# 13.1 American College of Rheumatology SLE Classification Criteria

The 1982 revised criteria for classification of systemic lupus erythematosus

| Criterion | Definition |
|---|---|
| 1. Malar rash | Fixed erythema, flat or raised, over the malar eminences, tending to spare the nasolabial folds |
| 2. Discoid rash | Erythematous raised patches with adherent keratotic scaling and follicular plugging; atrophic scarring may occur in older lesions |
| 3. Photosensitivity | Skin rash as a result of unusual reaction to sunlight, by patient history or physician observation |
| 4. Oral ulcers | Oral or nasopharyngeal ulceration, usually painless, observed by physician |
| 5. Arthritis | Nonerosive arthritis involving 2 or more peripheral joints, characterized by tenderness, swelling, or effusion |
| | <ul> <li>a) Pleuritisconvincing history of pleuritic pain or rubbing heard by a physician<br/>or evidence of pleural effusion</li> </ul> |
| 6. Serositis | OR |
| | b) Pericarditis-documented by ECG or rub or evidence of pericardial effusion |
| | a) Persistent proteinuria greater than 0.5 grams per day or grater than 3+ if quantitation not performed |
| 7. Renal disorder | OR |
| | b) Cellular castsmay be red cell, hemoglobin, granular, tubular, or mixed |
| | a) Seizuresin the absence of offending drugs or known metabolic derangements; e.g., uremia, ketoacidosis, or electrolyte imbalance |
| 8. Neurologic<br>disorder | OR |
| | b) Psychosisin the absence of offending drugs or known metabolic derangements, e.g., uremia, ketoacidosis, or electrolyte imbalance |
| | a) Hemolytic anemiawith reticulocytosis |
| | OR |
| | b) Leukopenialess than 4,000/mm<>3<> total on 2 or more occasions |
| 9. Hematologic | OR |
| disorder | c) Lymphopenialess than 1,500/mm<>3<> on 2 or more occasions |
| | OR |
| | d) Thrombocytopenialess than 100,000/mm<>3<> in the absence of offending drugs |
| 10. Immunologic | a) Positive LE cell preparation |

| | b) Anti-DNA: antibody to native DNA in abnormal titer |
|---|---|
| | OR |
| | c) Anti-Sm: presence of antibody to Sm nuclear antigen |
| | OR |
| | d) False positive serologic test for syphilis known to be positive for at least 6 months and confirmed by <i>Treponema pallidum</i> immobilization or fluorescent treponemal antibody absorption test |
| 11. Antinuclear<br>antibody | An abnormal titer of antinuclear antibody by immunofluorescence or an equivalent assay at any point in time and in the absence of drugs known to be associated with "drug-induced lupus" syndrome |

<sup>\*</sup> The proposed classification is based on 11 criteria. For the purpose of identifying patients in clinical studies, a person shall be said to have systemic lupus erythematosus if any 4 or more of the 11 criteria are present, serially or simultaneously, during any interval of observation.

Tan EM, Cohen AS, Fries JF, Masi AT, McShane DJ, Rothfield NF, et al. The 1982 revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum 1982; 25:1271---7.

### 13.2 Drug Formulations

### Cyclophosphamide

Other names:

Cytoxan, Neosar

Description:

2-bis (2-chloroethyl) amino tetrahydro-2H-1, 3, 2-

oxazaphosphorine-2-oxide monohydrate

Classification:

Alkylating agent

Action:

Causes prevention of cell division by forming adducts with

DNA

Metabolism:

Metabolized to active compounds by microsomal enzymes in

the liver. Excreted by the kidney in both the original form and

as metabolites.

Availability:

25 mg and 50 mg tablets (tablets cannot be split); 100 mg, 200 mg, 500 mg, 2000 mg vials Mead Johnson and Adria.

Storage:

Stable at room temperature indefinitely before reconstitution. After reconstitution, stable for 6 days upon refrigeration or for

24 hours at room temperature.

Administration:

Dissolved in 250 cc D5W and administered over 30-60 minutes IV. Must be aggressively hydrated before, during, and for 24 hours after cyclophosphamide. The rate of hydration required may not be tolerated in a patient with Jupu

hydration required may not be tolerated in a patient with lupus nephritis and in this case, bladder irrigation may need to be

substituted.

Side effects

Myelosuppression, leukopenia (nadir 8-14 days), hemorrhagic cystitis, syndrome of inappropriate secretion of antidiuretic hormone (SIADH), bladder carcinoma, cellular dysplasias, mucositis, rash, alopecia, anorexia, nausea, vomiting, sterile

phlebitis, rare pulmonary toxicity, teratogeneicity,

hemorrhagic, myocarditis, infertility, secondary leukemia; with

rapid IV push, oropharyngeal tingling, metallic taste,

headache, urticaria, facial swelling. Metabolic abnormalities following cyclophosphamide induced cell lysis can require dialysis in-patients with underlying renal insufficiency.

ATG (rabbit)

Other names: thymoglobulin

Classification: Biologic response modifier

Action: A rabbit polyclonal antibody to lymphocytes against human T-

lymphocytes. Exact mechanism of action is unknown.

07-22-2015

Availability:

50mg/ml (5 ml ample) vial.

Storage: Administration: Store ampules at 2-8 degrees centigrade.

Diluted in 250 NS and infused over 10 hours.

ATG (rabbit)
Side effects

Side effects of ATG are serum sickness and/or anaphylaxis: chills, arthralgias, headache, myalgias, nausea, vomiting, diarrhea, chest-pain, hypotension, dyspnea, pulmonary edema, abdominal pain. Other side effects include abnormal liver function tests (SGOT, SGPT) abnormal renal function,

and thrombocytopenia.

Rituximab

Other names:

Rituxan®

Classification:

Biologic response modifier

Action:

chimeric murine/human monoclonal antibody to the CD20 molecule on B-lymphocytes, The molecule is combined with Fc fragment of human IgG 1 kappa immunoglobulin containing murine light- and heavy-chain variable region sequence and human constant region sequences. Exact mechanism of

action is unknown.

Availability:

10mg/ml (10 ml and 50ml amples).

Storage:

protected from light at 2-8 degrees centigrade.

Administration:

Patients should be premedicated with 25mg diphenhydramine and 650mg of acetaminophen 30 minutes prior to the each rituximab infusion. The dose of 500 mg will be diluted in 500 cc 0.9%NS and infused per standard rituximab infusion guidelines (start at 50mg/h. If no reaction occurs, increase by 50mg/h every 30 minutes, to a maximum of 400mg/h.

Side effects

The most serious adverse reactions caused by rituximab include infusion reactions, mucocutaneous reactions, hypersensitivity reactions, cardiac arrhythmias and angina, and renal failure. The infusion reactions can be treated with slowing or interruption of the infusion and supportive care

(diphenhydramine, acetaminophen, IV satine or

vasopressors). Other reactions include:

nausea/vomiting/diarrhea, headache, myalgias, arthralgias.

cough, rhinitis, broncospasm, dyspnea, sinusitis,

lymphopenia, leukopenia, neutropenia, thrombocytopenia, anemia, abdominal pain, back pain, throat irritation, asthenia, infection. Reactivation of hepatitis B virus and progression to fulminant hepatitis has been reported in patients with negative hepatitis B surface antigen, but positive hepatitis B surface

antibody.

G-CSF

Other names: Filgrastim, Neupogen
Classification: Colony stimulating factor


G-CSF

Action: Stimulates the production, maturation, and activation of

neutrophils, G-CSF activates neutrophils to increase both their

migration and cytotoxicity.

Availability:

300 mcg and 480 mcg vials

Storage:

Stored in refrigerator

Administration:

Subcutaneous administration 5-15 mcg/kg/day

Side effects

Myalgias, headache, flu-like symptoms, fever, Bone pain in approximately 20% of patients, possible elevation of uric acid,

transaminases, and LDH.

#### 13.2 SF-36

# Short Form- 36 Health Survey (SF-36)

**INSTRUCTIONS:** The survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities.

Answer every question by marking the answer as indicated. If you are unsure about how to answer a question, please give the best answer you can.

| 1. | In general, would you say your health is: (circle one) | |
|---|---|---|
| | Excellent | 1 |
| | Very Good | 2 |
| | Good | 3 |
| | Fair | 4 |
| | Poor | 5 |
| 2. | COMPARED TO ONE YEAR AGO, how would you re NOW: (circle one) | ate your health in generat |
| | Much better now than one year ago | 1 |
| | Somewhat better now than one year ago | 2 |
| | About the same as one year ago | 3 |
| | Somewhat worse now than one year ago | 4 |
| | Much worse now than one year ago | 5 |

# 3. The following items are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

Circle one number on each item

| | ACTIVITIES | Yes,<br>Limited<br>A Lot | Yes,<br>Limited<br>A Little | No<br>Not<br>Limited<br>At All |
|---|---|---|---|---|
| a. | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports. | 1 | 2 | 3 |
| b. | Moderate activities, such as moving a table3 pushing a vacuum cleaner, bowling, or playing a | | 22 | 3 |
| c. | Lifting or carrying groceries. | 1 | 2 | 3 |
| d. | Climbing several flights of stairs. | | 2 | 3 |
| e. | Climbing one flight of stairs. | I | 2 | 3 |
| f. | Bending, kneeling, or stooping. | 1 | 2 | 3 |
| g. | Walking more than a mile. | | 2 | 3 |
| h. | Walking several blocks. | 1 | 2 | 3 |
| i. | Walking one block. | 1,5 | 2 | 3 |
| i. | Bathing or dressing yourself. | 1 | 2 | 3 |

| 4. | | During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of your physical health? |
|---|---|---|
| | | Circle one number on each line |
| | a. | Cut down on the amount of time you spent on work or 1 2 other activities. |
| | b. | Accomplished less than you would like. 1 2 |
| | c. | Were limited in the kind of work or other activities. 1 2 |
| | d. | Had difficulty performing the work or other activities 1 2 (for example, it took extra effort). |
| 5. | | During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of any emotional problems (such as feeling depressed or anxious)? Circle one number on each line. YES NO a. Cut down on the amount of time you spent on work or 1 2 other activities. b. Accomplished less than you would like. 1 2 c. Don't do work or other activities as carefully as usual. 1 2 |

| QF | groups? | Circle one |
|---|---|---|
| | Not at all | 1 |
| | Slightly | 2 |
| | Moderately | 3 |
| | Quite a bit | 4 |
| | Extremely | • |
| Ho | ow much bodily pain have you had during | g the past 4 weeks? |
| Ho | ow much bodily pain have you had during | g the past 4 weeks? Circle one |
| Но | ow much bodily pain have you had during | g the past 4 weeks? Circle one |
| Ho | ow much bodily pain have you had during | g the past 4 weeks? Circle one |
| Ho | NoneVery mild | circle one1 |
| Но | None | g the past 4 weeks? Circle one 2 3 |

| 8. | During the past 4 weeks, how much (including both work outside the ho | | | | | | nal wor<br>Circle o | |
|---|---|---|---|---|---|---|---|---|
| | Not at all | | | | | | 1 | |
| | Slightly | | ********** | | | 52 <i>9454</i> \$4446 | 2 | |
| | Moderately | | | | •••• | | 3 | |
| | Quite a bit | | | | | | .4 | |
| | Extremely | | ********** | | | | 5 | |
| 9. | These questions are about how you during the past 4 weeks. For each questiones closest to the way you have be the much of the time during the past 4 weeks. | uestio<br>een fe | n, plca<br>eling. | | the one | | r that | |
| | | the<br>Time | All of<br>of the<br>Time | Most<br>Bit of<br>Time | A<br>Good<br>of the<br>Time | Some<br>of the<br>Time | A<br>Little<br>of the<br>Time | None |
| a. D | Pid you feel full of pep? | 1 | 2 | 3 | 4 | 5 | 6 | |
| b. H | lave you been a very nervous person? | <u>l</u> | 2 | 3 | 4 | 5 | 6 | |
| | lave you felt so down in the dumps that othing could cheer you up? | 1 | 2 | 3 | 4 | 5 | 6 | |
| | lave you felt calm and peaceful? | | | | | | | |
| e. E | Did you have a lot of energy? | | 2 | 3 | 4 | 5 | 6 | |
| f. H | ave you felt downhearted and blue? | 1 | 2 | 3 | 4 | 5 | 6 | |
| g. Di | d you feel worn out? | 1 | 2 | 3, | 4 | 5 | 6 | |
| h. F | lave you been a happy person? | 1 | 2 | 3 | 4 | 5 | 6 | |
| i. D | id you feel tired? | | 2 | 3 | 4 | 5 | 6 | |

| 10. | During the past 4 weeks, how mucl problems interfered with your soci | | | | ıds, re | |
|---|---|---|---|---|---|---|
| | All of the time | | | 1 | | |
| | Most of the time | | | 2 | | |
| | Some of the time | *********** | ••••• | 3 | | |
| | A little of the time | | | 4 | | |
| | None of the time | | | 5 | | |
| 11. | How TRUE or FALSE is each of the | ne followit | ıg sta | atements for ye | ou? | |
| | (Circle one number on each line) | Definitely<br>True | Mo<br>True | • | Mostly<br>False | Definitely<br>False |
| a. | I seem to get sick a little easierthan other people | 1 | 2 | 3 | 4 | 5 |
| b. | I am healthy as anybody I know | ! | .2 | 3 | 4 | 5 |
| c. | I expect my health to get worse | 1 | 2 | 3 | 4 | 5 |
| d. | My health is excellent. | 1 | 2 | 3 | . 4 | 5 |
| I confi | rm that the information on this survey | is accurate | <b>.</b> | Patient's initials: | | Date: |
| | | | | Staff initials: | | Date: |
